CLINICAL TRIAL: NCT04595903
Title: Treatment of SARS-CoV-2 Virus Disease (COVID-19) in Humans With Hemopurifier® Device
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of eligible COVID-ICU patients
Sponsor: Aethlon Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AEMD-2020-02
Record Dates: First submitted 2020-10-08; First posted 2020-10-22 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: COVID-19
Keywords: Hemopurifier; SARS-CoV-2; COVID-19; exosomes; plasmapheresis
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This trial will evaluate the use of the Hemopurifier in patients with SARS-CoV-2 Virus Disease (COVID-19). The Hemopurifier is an extracorporeal device device that combines plasma filtration, size exclusion and affinity binding of mannosylated structures including enveloped viruses and exosomes. The study will evaluate whether the device is safe in COVID-19 patients along with clearing virus and improving outcomes in infected patients. Subjects will receive a four to six hour treatment with the Hemopurifier® extracorporeal therapy daily for up to four days until discontinued because of clinical improvement or deterioration or upon decision of the Principal Investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Hemopurifier® (Experimental): The Hemopurifier® will be placed within the extracorporeal circuit, all connections secured, treatment will utilize a blood pump at a flow rate of up to 200mL/min. The patients will be monitored for adverse events, device deficiencies and the development of hemodynamic instability. The treatment session will be for 4-6 hours once daily for 4 consecutive days.
  Interventions: Device: Hemopurifier

INTERVENTIONS:
Device: Hemopurifier — Hemopurifier treatments will be one four to six hour treatment session daily for up to 4 days

SUMMARY:
This is an Early Feasibility Study (EFS) investigating the use of the Hemopurifier® in the treatment of SARS-CoV-2 Virus Disease (COVID-19).

DETAILED DESCRIPTION:
Up to 40 ICU patients with severe or critical illness due to confirmed COVID-19 infection will be enrolled in up to 20 investigational sites. Patients will receive a four to six-hour treatment with the Hemopurifier® extracorporeal therapy daily for up to four days until discontinued because of clinical improvement or deterioration or upon the decision of the Principal Investigator. The patients will be monitored closely with vital signs and for hemodynamic stability. Patients will be followed for adverse events and device deficiencies. Blood work will be obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Laboratory diagnosis of COVID-19 infection with any of the following disease characteristics:

   i. Early acute lung injury (ALI)/early acute respiratory distress syndrome (ARDS) ii. Severe disease, defined as:
   * dyspnea,
   * respiratory frequency ≥ 30/min,
   * blood oxygen saturation ≤ 93%,,
   * partial pressure of arterial oxygen to fraction of inspired oxygen ratio of <300 and/or
   * lung infiltrates >50% within 24 to 48 hours; iii. Life-threatening disease, defined as:

     1. respiratory failure,
     2. septic shock, and/or
     3. multiple organ dysfunction or failure.
2. Admission to the ICU or area of the hospital repurposed to function as an ICU for surge capacity management
3. Subject has maintained a MAP of > or = 65 without an increased dose of vasopressors for at least 2 hours and has clinical evidence of adequate volume status per investigative site criteria
4. Informed consent from the patient or legally authorized representative
5. Age > 18

Exclusion Criteria:

1. Stroke (known or suspected) within the last 3 months.
2. Severe congestive heart failure (NYHA III and IV classes).
3. Biopsy proven cancer not in remission.
4. Acute (an international normalized ratio (INR) of greater than 1.5, and any degree of mental alteration (encephalopathy) in a patient without preexisting cirrhosis and with an illness of less than 26weeks' duration or chronic (Child Pugh C) liver disease.
5. Known pre-existing non-COVID-19 related hypercoagulability or other coagulopathy
6. Terminal illness with a life expectancy of < 28 days or for whom a decision of withdrawal of care is in place or imminently anticipated or patients who have received prior extracorporeal therapy and had persistent, unstable hypotension.
7. Patients with known hypersensitivity to any component of the Hemopurifier.
8. Advance directive indicating to withhold life-sustaining treatment (except Cardiopulmonary Resuscitation).
9. Contraindications to extracorporeal blood purification therapy such as:

   i. Clinically relevant bleeding disorder, ii. Contraindication to anti-coagulation, iii. Pregnancy, iv. Inability to establish functional vascular access, v. Participation in another competing investigational drug, device or vaccine trial vi. Administration of an angiotensin converting enzyme (ACE) inhibitor in the previous 14 days. vii. Platelet count < 50,000 cells/microliter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | Day 1 (Date of Consent) to Day 28
  Safety and tolerability
Incidence of device related adverse events | Day 1 (Date of Consent) to Day 14
  Safety and tolerability with adverse event graded at 2 or higher
Incidence of serious adverse events | Day 1 (Date of Consent) to Day 28
  Safety and tolerability

SECONDARY OUTCOMES:
Length if Stay in ICU | Day 1 (Date of Consent) to Day 28
  Length of ICU stay in days
In-hospital mortality | Day 1 (Date of Consent) to Day 28
  Number of deaths during hospitalization
Days free of ventilatory dependency | Day 1 (Date of Consent) to Day 28
  Number of days without ventilatory support
Vasopressor-free days | Day 1 (Date of Consent) to Day 28
  Number of days without vasopressor support
Sequential Organ Failure Assessment (SOFA) | Before first daily filter treatment and after the last daily filter treatment (i.e. 4 days or more)
  SOFA scoring system predicts the clinical outcome of critically ill patients.
Acute Physiology and Chronic Health Evaluation (APACHE) | Before first daily filter treatment and after the last daily filter treatment (i.e. 4 days or more)
  Measures the severity of disease for adult patients admitted to an ICU
SARS CoV-2 RNA levels in plasma and nasopharyngeal samples | Before each filter treatment, every 2 hours during filter treatment and immediately after filter discontinued
  Measures viral exposure and levels of circulating virus
Total lymphocyte count | Before first daily filter treatment and after the last daily filter treatment (i.e. at 4 days or more)
  Measurement of lymphocytes as there seems to be a correlation with the disease severity and lymphopenia.
C-reactive protein (CRP), IL-1, IL-6, and TNF alpha Tests | Before first daily filter treatment and after the last daily filter treatment (i.e. at 4 days or more)
  Measurement of inflammatory marker levels play a role in systemic vasculitis and cytokine mediated coagulation disorders as the principal actors of multi organ failure in patients with severe COVID-19 complication.
D-dimer | Before first daily filter treatment and after the last daily filter treatment (i.e. at 4 days or more)
  Measurement of D-dimer levels as levels are elevated in patients with COVID-19 and correlate with disease severity, are a reliable prognostic marker for in-hospital mortality.
Troponin-T | Before first daily filter treatment and after the last daily filter treatment (i.e. at 4 days or more)
  Measurement of Troponin-T as high levels of troponin is found in COVID-19 patients.
Evaluation of SARS-CoV-2 RNA levels post-treatment Hemopurifier cartridges | Until study completion, 1 week or for the duration of ICU admission
  Measures the levels of SARS-CoV-2 RNA captured in the filter
Evaluation of viral particle load post-treatment Hemopurifier cartridges | Until study completion, 1 week or for the duration of ICU admission
  Measures the levels of viral particles captured in the filter

CONTACTS AND LOCATIONS:
Overall Officials: Steven LaRosa, MD, Study Director — Aethlon Medical Inc.
Locations (9):
- United States (9):
  - Hoag Hospital - Irvine, Irvine, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - UC Davis Health System, Sacramento, California
  - University of Miami Hospital, Miami, Florida
  - LSU Health Sciences Center, Shreveport, Louisiana
  - Cooper University Hospital, Camden, New Jersey
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Valley Baptist Medical Center, Harlingen, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amundson DE, Shah US, de Necochea-Campion R, Jacobs M, LaRosa SP, Fisher CJ Jr. Removal of COVID-19 Spike Protein, Whole Virus, Exosomes, and Exosomal MicroRNAs by the Hemopurifier(R) Lectin-Affinity Cartridge in Critically Ill Patients With COVID-19 Infection. Front Med (Lausanne). 2021 Oct 8;8:744141. doi: 10.3389/fmed.2021.744141. eCollection 2021. PMID 34692735
- [Background] Gooldy M, Roux CM, LaRosa SP, Spaulding N, Fisher CJ Jr. Removal of clinically relevant SARS-CoV-2 variants by an affinity resin containing Galanthus nivalis agglutinin. PLoS One. 2022 Jul 28;17(7):e0272377. doi: 10.1371/journal.pone.0272377. eCollection 2022. PMID 35901224
- See also: Website — https://www.frontiersin.org/articles/10.3389/fmed.2021.744141/full
- See also: Website — https://www.biorxiv.org/content/10.1101/2022.04.27.489436v1.full